CLINICAL TRIAL: NCT03425734
Title: The Effect of Dexmedetomidine on Kidney Perfusion in Paediatric Patients Undergoing Open Heart Surgery Guided by Near Infrared Spectroscopy: Randomized Controlled Study
Brief Title: The Effect of Dexmedetomidine on Kidney Perfusion in Paediatric Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mai Madkour (Other)
Responsible Party: Sponsor-Investigator, Mai Madkour, lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N19234
Record Dates: First submitted 2018-01-17; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D group (Experimental): The drug will be prepared in 50 ml saline 0.5 ml DEX (100mc/ml +49.5 cc saline 1ml=1mg), and the dose will be calculated according to body weight.
  Interventions: Drug: Dexmedetomidine
- S group (Experimental): 50 ml saline
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The drug will be prepared in 50 ml saline 0.5 ml DEX (100mc/ml +49.5 cc saline 1ml=1mg), and the dose will be calculated according to body weight.

SUMMARY:
I. Study design: open/ blinded randomized, controlled study.

II. Study setting and location:

The study will be conducted in Abul Reesh Paediatric Hospital Faculty of Medicine /Cairo University from 2016-2018.

III. Study population:

This controlled open/blinded labelled randomized study is designed to include 40 children of both sexes scheduled for open-heart surgery for total correction of congenital heart diseases.

IV. Eligibility Criteria:

Inclusion criteria;

1. Paediatric patients of age group ranging from 6 months to 12 years .
2. Patients with complex congenital heart disease undergoing open heart surgery for total correction of the cardiac anomaly using cardiopulmonary bypass.

Exclusion criteria;

* Age less than 6 months or more than12 years.
* Significant ventricular dysfunction (Ejection fraction < 40%).
* Patients with pre-existing CNS disorders e.g.: seizures.
* Patients with abnormal liver functions.
* Pre-operative creatinine level >1.2 mg /dl.
* Patients with history of diabetes mellitus.
* Patients receiving NSAID for any reason. Study Protocol; The patients will be pre-medicated by atropine 0.01mg/kg, ketamine 0.03mg/kg and midazolam 0.02mg/kg IM, 30 minutes before induction of anesthesia. Standard ASA monitors, including electrocardiogram (ECG), pulse oximetry (Spo2), and non-invasive blood pressure cuff, and INVOS somatic oximeter probes will be placed on the renal area (on the back to the right or to the left from T10 to l2) will be placed on the patients before induction of anesthesia.

Anesthetic technique will be standardized for all the patients in the form of inhalational induction using sevoflurane 6% in a mixture of oxygen and air (1:1) to be followed by placement of peripheral intravenous cannula. Intubation will be facilitated by pancuronium 0.01 mg/kg IV and ventilation will be controlled using pressure mode aiming to maintain PCO2 between (30-35 mmHg). Anesthesia will be maintained by mixture of 2% sevoflurane in 1:1 oxygen: air till time of CPB.

A standard CPB technique will be used in all patients. Before aortic cannulation, patients will receive IV heparin 400 U.kg-1 aiming to produce ACT value > 400 sec. A membrane oxygenator (minimax plus ;Medtronics Inc.,Anaheim,CA) will be used during CPB. Priming solution in the form of isotonic saline solution supplemented with heparin added to fresh whole blood in appropriate amounts to achieve a hematocrit 20-25% during CPB will be used. Furosemide in a dose of 1mg .kg-1.min-1 will be given to all patients. Venting of left heart will be performed with a left atrial vent inserted through a small incision at the inter-atrial septum . Anesthesia during CPB will be given by Sevoflurane administrated via a vaporizer inserted into the oxygenator gas supply with a constant gas flow 3 liter.min-1. A non-pulsatile roller pump (model10.10.00;Stocket instruments ;Munich, Germany) will be used and the pump flow will be adjusted at 2.4 to 2.6 L/min /m2 during the normothermic period targeting mean arterial blood pressure between 40 and 60 mmHg. If the MAP will fall below 40 mmHg despite full perfusion pressure, a bolus dose of 0.01-0.1 ng /Kg phenylephrine will be given. If MAP increased above 60 mmHg, a continuous infusion of nitroglycerin at a dose of 1-2 µg.kg.min-1will be given.

After application of aortic cross clamp and administration of cold cardioplegia solution (Saint Thomas cardioplegic solution, 20ml/Kg to be followed by doses of 10ml/Kg every 20 min.), time will be allowed to develop a stable level of perfusion pressure and moderate hypothermia (28°C-32°C).

These variables will be kept constant for at least 10 minutes after initiation of full flow CPB and initiation of the study sequence. Thereafter, patients will be randomely allocated to DEX group (Group D n=20) receiving dexmedetomidine in a dose of 3 mcg/kg over 10 minutes to be followed by an infusion of 1 mcg/kg/hr to be continued until the first 6 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* children 6m to 12 years complex congenital heart disease

Exclusion Criteria:

* signifiacnt ventricular dysfunction pre-existing CNS disorders

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-05-20 (Estimated); Study Completion 2018-07-20 (Estimated)

PRIMARY OUTCOMES:
renal regional oxygen saturation | 24 hours
  compares regional renal oxygen saturation measured by invos with and without dexmedetomidine infusion

SECONDARY OUTCOMES:
urine output | 24 hours
  measured across the day by urinary catheter

CONTACTS AND LOCATIONS:
Overall Officials: A Shash, Study Chair — Anesthesia Dep
Locations (1):
- Pediatric University Hospitals, Cairo, Outside US and Canada, Egypt

IPD SHARING:
Plan to Share IPD: No